CLINICAL TRIAL: NCT01689675
Title: Pain Management Following Musculoskeletal Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: NA_00049927; 1R01AR054009-01A1 (NIH)
Record Dates: First submitted 2012-09-07; First posted 2012-09-21 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Musculoskeletal Strain; Musculoskeletal Sprain; Injury of Musculoskeletal System
Keywords: musculoskeletal; pain; pain management; computer based intervention
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer based pain management (Experimental): The computer-based self-management program (CBSM) intervention will be administered over 8 sessions during the average 4 week period patients are receiving their standard on-site rehabilitation care. Patients will come to the center to receive their standard care and then interact with the computer for the 25-30 minute CBSM intervention. The primary goals of treatment include developing skills for managing acute injury and related pain including: reducing fear avoidance beliefs and catastrophizing, improving mood, increasing perceptions of control and self-efficacy, maintaining activity and reducing pain. Skills are presented and modeled by computer-based video during sessions, audio will be used to explain models and teach skills such as relaxation training.
  Interventions: Behavioral: Computer based pain management
- Education control (Active Comparator): The computer exposure will be administered over 8 sessions during the average 4-week period patients are receiving their standard on-site rehabilitation care. Patients will come to the center to receive their standard care and then interact with the computer for the 25-30 minute control condition. The primary goal of this condition is to provide a control for computer exposure. Briefly, the first session will concentrate on establishing the patient's ability to interact with the computer. The materials will provide general education regarding the injury and methods for preventing re-injury. This condition will not provide teaching and practice of specific pain management and coping management skills. This control computer education activity will equalize the computer exposure of the two groups and the duration of time devoted to injury care.
  Interventions: Behavioral: Computer based pain management

INTERVENTIONS:
Behavioral: Computer based pain management

SUMMARY:
Musculoskeletal sprain/strain injuries and disorders (MSID) have a major impact on health, quality of life and societal productivity. Early intervention for pain following acute MSIDs may prevent secondary complications of chronic pain, disability, reduced quality of life or lost productivity. The investigators goal is to evaluate the efficacy of a computer-based self-management intervention for reducing pain and improving function in persons treated in on-site physical rehabilitation centers.

The specific aims are:1) evaluate the efficacy of a computer-based self-management intervention in reducing pain and self-efficacy and function in high risk MSID patients; 2) determine long term impact during a six month follow-up period; and 3) determine whether reductions of pain and improved function translate into reductions in lost work time days away from work, restricted work days, worker's compensation costs and re-injury rates during the 6 month follow-up.

Persons with sprain/strain injuries at risk for poor pain control will randomized to either: 1) control condition - standard care in the rehabilitation center plus computer exposure or 2) standard care plus computer-based self-management pain intervention. Assessment will be at baseline, treatment completion, 3 and 6 months. The primary outcome measures are self-efficacy, pain and physical/psychosocial functioning and secondary outcome measures are days away from work, restricted work days worker's compensation costs and re-injury rates. The investigation will also provide unique and valuable information regarding patients acceptance and use of computer-based interventions following acute injury. By establishing the utility and efficacy of computer-based pain management interventions for MSID the investigators have the potential to improve the health and quality of life of persons with injuries, improve productivity and develop new methods for health care delivery.

DETAILED DESCRIPTION:
The proposed study will use a 2 group randomized controlled clinical trial design. The two groups are: 1) standard care in the rehabilitation center with control computer exposure (SCCE) and 2) standard care plus computer-based self-management pain (CBSM) intervention. The study will examine the short- and long-term effects of these interventions on pain and physical and psychosocial functioning and productivity (DAW, RWD, WC costs and re-injury) in 200 completing patients with strain/sprain MSID. Outcome data will be collected at baseline, after treatment, and at 3 and 6 month follow-up. All outcome assessments will be administered by computer.

Pain Management Following Musculoskeletal Injury Study. The study is comprised of two phases: Phase I Planning/Development and Phase II Intervention.

During Phase I Planning/Development, the study investigators 1) identified technology partner to aid in computerization of intervention; 2) identified sites for study implementation; 3) developed consent forms and tracking procedures; 4) developed computer based self-management (CBSM) pain intervention; 5) developed computer based educational materials for the control condition; 6) beta tested intervention materials; 7) developed recruitment materials; 8) developed outcome assessment procedures measures.

During Phase II Intervention, the study investigators will 1)complete IRB review at each of the study sites; 2) train study personnel, and upon approval from each of the IRBs; 3) initiation of study subject recruitment and intervention. Phase II will begin June 2011 and be completed by June 2013.

During Phase II a total of 200 patients will be enrolled in the study.

Control Group Individuals with acute MSID, in the employers with on-site rehabilitation centers, are initially seen by the plant medical office and, if appropriate, referred for rehabilitation services. Patients are given an initial evaluation by the treating physical or occupational therapist and a treatment plan is implemented. The typical patient is seen for an average of approximately 9 visits over a four-week period. However, patients can be seen as long as indicated. SCCE is seen as the appropriate control condition for several reasons. First, denying patients care is not ethically appropriate. Second, this is type of rehabilitation and injury education is the care typically received by acute MSID patients and is the current standard of practice. Currently the education is provided in written brochures and handouts. The addition of computer interaction for presenting this education controls for threats related to differential time spent in treatment and the novelty of computer supplement to care. The computer exposure will be administered over 8 sessions during the average 4-week period patients are receiving their standard on-site rehabilitation care. Patients will come to the center to receive their standard care and then interact with the computer for the 25-30 minute control condition. The primary goal of this condition is to provide a control for computer exposure. Briefly, the first session will concentrate on establishing the patient's ability to interact with the computer. The materials will provide general education regarding the injury and methods for preventing re-injury. This condition will not provide teaching and practice of specific pain management and coping management skills. This control computer education activity will equalize the computer exposure of the two groups and the duration of time devoted to injury care.

Intervention Group: Will receive the same medical care and physical therapy treatment as the control group. In addition the computer-based self-management program (CBSM) intervention will be administered over 8 sessions during the average 4 week period patients are receiving their standard on-site rehabilitation care. Patients will come to the center to receive their standard care and then interact with the computer for the 25-30 minute CBSM intervention. The primary goals of treatment include developing skills for managing acute injury and related pain including: reducing fear avoidance beliefs and catastrophizing, improving mood, increasing perceptions of control and self-efficacy, maintaining activity and reducing pain. The intervention materials are based on the investigators work in the a self-management program for persons with limb loss and those shown effective in other secondary prevention studies in MSID, specifically the Pain Disability Prevention Program (PDPP) develop by Sullivan. While the PDPP has been evaluated on persons who have been out of work for six weeks or more and this study targets individuals who are more recently injured, the content of the intervention is appropriate for the study population. Each session focuses on specific topics and sets of skills. Skills are presented and modeled by computer-based video during sessions, audio will be used to explain models and teach skills such as relaxation training. This will supplement any written materials and minimize the need for reading. Patients are instructed to practice and apply skills between sessions. Patients will also be given specific feedback about their progress in working through the CBSM modules. As all CBSM takes place within the on-site rehabilitation center, staff are available to provide assistance if necessary. The sessions initially focus on pain, which is a primary motivator to the patient, expand the focus to cognitive and emotional factors related to pain and disability and finally move to increasing activity. A home activity will be assigned at completion of the session. The home activity will be printed out for the patient to take home and will be available to the participant through the study website from remote locations. The study intervention and home activities will be refined using focus group and pilot testing methods.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older
2. Musculoskeletal sprain/strain injury
3. pain level greater or equal to 5
4. English speaking

Exclusion Criteria:

1. Age < 18
2. non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain | 3 month followup
  Pain will be measured using the Brief Pain Inventory, which includes 4 pain items assessing current, worst, least, and average pain (0-no pain to 10-as bad as you can imagine) during the past week. This scale has excellent reliability and validity in a wide variety of acute and chronically painful conditions. In addition to measuring pain severity, 10 items measure pain-related interference in daily activities (0-does not interfere to 10-completely interferes) which also shows excellent reliability and validity in a wide variety of acute and chronically painful conditions.
Physical and Psychosocial Function | 3 month followup
  The SF-12 was designed for use in clinical practice and research, health policy evaluations, and general population surveys. The SF-12 includes items that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. A total score and two subscales scores are calculated -physical function and psychosocial function. The survey was constructed for self-administration by persons 14 years of age and older, and for administration by a trained interviewer, self-report, or by telephone.

SECONDARY OUTCOMES:
Work Productivity | 3 month followup
  Work productivity will be measured by the number of days away from work, restricted work days, and Worker's compensation costs related to this incident of care. Due to the lost productivity and worker compensation cost associated with MSID, it is critical to include these measures in the outcome analyses 10. In addition, the number of re-injuries that occur following treatment will also be included as an outcome measure. These data are available through contacting Worker's Compensation intermediary. We have experience accessing, manipulating and analyzing these data for previous program evaluation cost benefit analyses.

OTHER OUTCOMES:
Catastrophizing | 3 month followup
  The Pain Catastrophizing Scale will be used to measure catastrophic thinking related to pain. Respondents rate the frequency with which they experience 13 different thoughts and feelings related to pain. The scale has been shown to be reliable (alpha =.87) and has been associated with pain levels, self-reported disability and employment status.
Self-Efficacy | 3 month followup
  There is evidence that enhancement of perceived self- efficacy may mediate pain control and improved psychosocial functioning in persons who participate in self-management intervention. Self-efficacy for pain management will be measured using the Pain Self-Efficacy scale which includes subscales that measure self-efficacy for pain management, self-efficacy for coping with symptoms, and self-efficacy for physical function.
Fear-avoidance beliefs | 3 month followup
  This variable will be measured with 2 questionnaires: 1) The Tampa Scale of Kinesiophobia (TSK), which has been shown to be a relevant measure of fear of movement/activity; 2) A modified form of the Fear-Avoidance Behavior Questionnaire that contains four items from the physical activity scales. These measures have both been associated with long term pain and work disability in acutely injured individuals.
Utility and Use of Intervention Materials | 4 weeks after starting treatment
  The use of computers for delivery of the intervention allows for ongoing monitoring of intervention activity materials. Quantitative metrics will be collected as part of the intervention including sessions attended, the amount of the program completed in each session, and utilization of Support Services (time on bulletin board and number of postings). Utilization of the website containing the intervention, Support Service and assessment materials will be evaluated for (1) the effectiveness with which users can accomplish tasks; (2) the speed with which users can find the information they are seeking and navigate through the elements of the prototype session; (3) the paths users take to complete a task; and 4) users' satisfaction level using the interactive tools. Qualitative data to be collected includes: user comments, concerns, frustrations, and suggestions.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Wegener, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee